CLINICAL TRIAL: NCT01203566
Title: A Double-blinded Randomised Controlled Trial of Laparoendoscopic Single-site Access (LESS) Versus Conventional Three-port Appendicectomy.
Brief Title: A Randomised Controlled Trial on LESS Versus Conventional Laparoscopic Appendicectomy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Anthony Yuen Bun Teoh, Department of Surgery, Chinese University of Hong Kong, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CREC 2009.347
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2010-09

CONDITIONS: Appendicitis
Keywords: Single incision laparoscopic surgery; Single site access laparoscopic surgery; SILS; Single-port access; Laparoendoscopic single site surgery; Appendectomy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional 3-port laparoscopic appendectomy (Active Comparator): Laparoscopic appendectomy will be performed with the standard 3-port technique. The laparoscope is introduced via a 10mm subumbilical port. Dissection will be performed with a 5mm LLQ port and a 5mm RLQ port. Exploratory laparoscopy was first carried out to locate the appendix and to rule out other pathologies. The mesoappendix will be divided with the ultrasonic dissector (Sonosurg, Olympus surgical, Tokyo, Japan). The appendix will be ligated between two polydioxanone suture loops. The specimen will be delivered within a plastic bag via the subumbilical port. Purulent fluid will be irrigated and suctioned from the subhepatic space, right lower quadrant and the pelvis if present. Fascial defects will be closed with 2-O polydioxanone sutures and skin closed with 4-O absorbable subcuticular sutures. A pelvic drain (12Fr) will be inserted in cases of abscesses or gangrene.
  Interventions: Procedure: Conventional 3-port laparoscopic appendectomy
- LESS appendectomy (Active Comparator): Two 5 mm ports and a 10mm port will be inserted through a 13mm transumbilical incision. Exploratory laparoscopy was first carried out to locate the appendix and to rule out other pathologies. Retraction of the appendix would be performed with a flexible curved forceps. The mesoappendix will be divided with the ultrasonic dissector (Sonosurg, Olympus surgical, Tokyo, Japan). The appendix will be ligated between two polydioxanone suture loops. The specimen will be delivered within a plastic bag via the subumbilical port. Purulent fluid will be irrigated and suctioned from the subhepatic space, right lower quadrant and the pelvis if present. Fascial defects will be closed with 2-O polydioxanone sutures and skin closed with 4-O absorbable subcuticular sutures. A pelvic drain (12Fr) will be inserted in cases of abscesses or gangrene.
  Interventions: Procedure: LESS appendectomy

INTERVENTIONS:
Procedure: LESS appendectomy — See under arms description
  Arms: LESS appendectomy
Procedure: Conventional 3-port laparoscopic appendectomy — See under arms description
  Arms: Conventional 3-port laparoscopic appendectomy

SUMMARY:
LESS laparoscopic appendectomy is associated with less pain than conventional 3-port laparoscopic appendectomy.

DETAILED DESCRIPTION:
Since the original description in the 1970's, the laparoscopic approach to management of surgical diseases has gained widespread acceptance. It has been shown to be associated with decreased wound pain, analgesic requirements, hospital stay and allows improved cosmesis and quality of life without significantly increasing the risks of morbidities and mortalities. With continued improvements in technology, however, efforts to reduce the number of abdomen wounds in an attempt to further decrease pain, improve cosmesis and outcomes are underway. Natural Orifices Transluminal Endoscopic Surgery (NOTES) has received widespread attention in both the medical field as well as the general public. However, there are still a multitude of problems that needs to be solved before the technique can be broadly applied to human subjects [7]. On the other hand, a renewed interest in single incision laparoscopic surgeries is emerging. The approach has been shown to be safe and feasible in our experience as well as the others. It also has the potential to further decrease the surgical trauma induced to the patient and to improve cosmesis.

Since laparoscopic appendicectomy is one of the most basic procedures in laparoscopic surgery, it is an appropriate model for initial evaluation of single incision laparoscopic surgery. Our unit has already performed 20 cases of single site access laparoscopic appendicectomy (SSALA) and so far, the results have been encouraging (data pending publication). All the patients in the series had their procedures completed with a single incision. None of the patients suffered from adverse events and all had resumption of oral diet by day 1 and were discharged on day 2 post-operatively. However, whether the approach is more beneficial as compared to conventional three-port laparoscopic appendicectomy is still uncertain.

Hence, the aim of the current study is to compare the approach of SSALA to conventional three-port laparoscopic appendicectomy in reducing surgical trauma and improving cosmesis to the patient.

ELIGIBILITY:
Inclusion Criteria:

* History of right lower quadrant pain or periumbilical pain migrating to the right lower quadrant
* Fever ≥ 38°C and/or WCC > 10 X 103 cells per mL,
* Right lower quadrant guarding, and tenderness on physical examination.
* All patients included were 18-75 years old.

Exclusion Criteria:

* Patients are excluded if the diagnosis of appendicitis is not clinically established (symptoms attributable to urinary or gynaecological problems).
* History of symptoms > 5 days and/or a palpable mass in the right lower quadrant, suggesting an appendiceal abscess treated with antibiotics and possible percutaneous drainage.
* Patients with the following conditions are also excluded: history of cirrhosis and coagulation disorders, generalized peritonitis, shock on admission, previous abdominal surgery, ascites, suspected or proven malignancy, contraindication to general anesthesia (severe cardiac and/or pulmonary disease), inability to give informed consent due to mental disability, and pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Overall pain score experienced by the patient within the last 24 hrs using the visual analogue scale | 1st post-operative day
  The main outcome is the overall pain score (measured as the most severe pain experienced within the last 24 hrs using the visual analogue scale) experienced by the patient after the operation

SECONDARY OUTCOMES:
Conversion | 24 hours
  defined by the use of incisions and/or trocars in addition to the ones described in the Methods section, or the need to perform an open procedure
Operative time | 24 hours
  defined as the amount of time to perform the operation from skin-incision to application of the dressing.
Wound infection | 14 days
  defined as presence of skin erythema, discharge and a positive culture
Deep space infection | 30 days
  defined as the need for reoperation, readmission, or percutaneous drainage of a deep (organ space) infection within 30 days of surgery.
activity score | 14 days
  defined by a composite score including 4 items using a five point scale: lying in bed, getting out of chair or bed, walking on level ground and climbing stairs [1. no difficulty; 2. a little difficult; 3. some difficulty; 4. a lot of difficulty; 5. not able to perform.]
Satisfaction score | 14 days
  Overall satisfaction of the procedure by the patient measured with the visual analogue scale
Cosmesis score | 14 days
  defined as the score given by the patient on the overall cosmesis of the wound measured by the visual analogue scale
quality of life | 14 days
  measured by the gastrointestinal quality of life index (GIQLI) and SF-36 at 2-weeks follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Y Teoh, FRCSEd (Gen), Principal Investigator — Chinese University of Hong Kong
Locations (2):
- China (2):
  - Deparment of Surgery, North District Hospital, Sheung Shui, Hong Kong
  - Department of Surgery, Prince of Wales Hospital, Shatin, Hong Kong

REFERENCES:
- [Background] Pappalepore N, Tursini S, Marino N, Lisi G, Lelli Chiesa P. Transumbilical laparoscopic-assisted appendectomy (TULAA): a safe and useful alternative for uncomplicated appendicitis. Eur J Pediatr Surg. 2002 Dec;12(6):383-6. doi: 10.1055/s-2002-36846. PMID 12548490
- [Background] Hong TH, Kim HL, Lee YS, Kim JJ, Lee KH, You YK, Oh SJ, Park SM. Transumbilical single-port laparoscopic appendectomy (TUSPLA): scarless intracorporeal appendectomy. J Laparoendosc Adv Surg Tech A. 2009 Feb;19(1):75-8. doi: 10.1089/lap.2008.0338. PMID 19196084
- [Background] Chow A, Purkayastha S, Paraskeva P. Appendicectomy and cholecystectomy using single-incision laparoscopic surgery (SILS): the first UK experience. Surg Innov. 2009 Sep;16(3):211-7. doi: 10.1177/1553350609344413. Epub 2009 Aug 31. PMID 19723692
- [Derived] Teoh AY, Chiu PW, Wong TC, Poon MC, Wong SK, Leong HT, Lai PB, Ng EK. A double-blinded randomized controlled trial of laparoendoscopic single-site access versus conventional 3-port appendectomy. Ann Surg. 2012 Dec;256(6):909-14. doi: 10.1097/SLA.0b013e3182765fcf. PMID 23154391